CLINICAL TRIAL: NCT05669079
Title: Decitabine and Umbilical Cord Blood for Poor Graft Function Post Allogenic Hematopoietic Stem Cell Transplantation
Brief Title: Decitabine and Umbilical Cord Blood for Poor Graft Function Post Allo-HSCT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2022-12-15
Record Dates: First submitted 2022-12-19; First posted 2022-12-30 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2022-12

CONDITIONS: Poor Graft Function
MeSH Terms: interventions — Decitabine; Granulocyte Colony-Stimulating Factor; Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): decitabine (Chia Tai Tianqing Pharma) 15 mg/m2 daily intravenously for consecutive 3 days (day 1 to day 3), combined with umbilical cord blood infusion (day 8)
  Interventions: Drug: decitabine; Biological: umbilical cord blood; Drug: Granulocyte-colony stimulating factor; Drug: Recombinant human thrombopoietin / thrombopoietin receptor agonist; Drug: Recombinant human erythropoietin
- Arm B (Active Comparator): Supportive therapy: G-CSF for patients with absolute neutrophil count ≤ 1.5 × 109/L, rhTPO/TPO-R with platelet count ≤ 30 × 109/L, EPO with hemoglobin ≤ 85g/L.
  Interventions: Drug: Granulocyte-colony stimulating factor; Drug: Recombinant human thrombopoietin / thrombopoietin receptor agonist; Drug: Recombinant human erythropoietin

INTERVENTIONS:
Drug: decitabine — 15 mg/m2 daily intravenously for consecutive 3 days
  Other Names: Dec
  Arms: Arm A
Biological: umbilical cord blood — MNC ≥ 3*108 cells; HLA compatibility ≥ 5/6
  Other Names: UCB
  Arms: Arm A
Drug: Granulocyte-colony stimulating factor — Granulocyte-colony stimulating factor will be used when absolute neutrophil count ≤ 1.5 × 109/L
  Other Names: G-CSF
Drug: Recombinant human thrombopoietin / thrombopoietin receptor agonist — Recombinant human thrombopoietin or thrombopoietin receptor agonist will be used when platelet count ≤ 30 × 109/L
  Other Names: rhTPO/TPO-RA
Drug: Recombinant human erythropoietin — Recombinant human erythropoietin will be used when hemoglobin ≤ 85 g/L
  Other Names: EPO

SUMMARY:
This randomized trial aimed at validating the efficacy and safety of low-dose decitabine, together with umbilical cord blood in PGF post allo-HSCT patients.

DETAILED DESCRIPTION:
Poor graft function (PGF), defined by the presence of multilineage cytopenias in the presence of 100% donor chimerism, is a serious complication of allogeneic stem cell transplant (allo-HSCT). Emerging evidence demonstrates that the inadequate stem cells infusion, bone marrow microenvironment and immune dysregulation play a crucial role in maintaining and regulating hematopoiesis. Current therapies remain debatable, including selected CD34+ cells infusion, mesenchymal stromal cells infusion, prophylactic N-acetyl cysteine administration, etc. Thereafter, the investigators conduct a randomized trial aiming at validating the efficacy and safety of low-dose decitabine, together with umbilical cord blood in PGF post allo-HSCT patients.

Patients were eligible if they were diagnosed as PGF at day 28 post-HSCT or later. PGF was defined as two or three cytopenias, absolute neutrophil count ≤ 1.5 × 109/L, platelet count ≤ 30 × 109/L, hemoglobin ≤ 85g/L, lasting for more than 14 consecutive weeks, in the presence of full donor chimerism and primary disease in remission without severe graft-versus- host disease (GVHD) and relapse.

Patients with the following conditions or diagnoses were excluded: allergic to decitabine or any components of frozen preservation of umbilical cord blood; active infections; uncontrolled GVHD; severe organ dysfunction; relapse of underlying malignancies; graft failure. Patients were also excluded if they had received decitabine or participated in other clinical trials within one month before screening.

Hematological improvement is defined as recovery of two or three blood lineages: absolute neutrophil count>1.5 × 109/L, platelet count>30 × 109/L, hemoglobin>85g/L, without G-CSF, red blood cell or platelet infusion.

Hematological response is defined as recovery of three blood lineages: absolute neutrophil count>2.5 × 109/L, platelet count>60 × 109/L, hemoglobin>100g/L, without G-CSF, red blood cell or platelet infusion.

No response: failed to achieve hematological improvement or response.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as PGF at day 28 post-HSCT or later. PGF was defined as two or three cytopenias, absolute neutrophil count ≤ 1.5 × 109/L, platelet count ≤ 30 × 109/L, hemoglobin ≤ 85g/L, lasting for more than 2 consecutive weeks;
2. Full donor chimerism;
3. Primary disease in remission;
4. No severe GVHD and relapse.

Exclusion Criteria:

1. Allergic to decitabine or any components of frozen preservation of umbilical cord blood;
2. Active infections;
3. Uncontrolled GVHD;
4. Severe organ dysfunction;
5. Relapse of underlying malignancies;
6. Graft failure;
7. Received decitabine or participated in other clinical trials within one month before screening.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The treatment response | day +28
  The rate of hematological improvement and hematological response of 2 arms
Survival | 1 year
  The rate of overall survival

SECONDARY OUTCOMES:
Bone marrow recovery | day +28
  Number of participants with granulopoiesis, erythropoiesis and megakaryopoiesis recovery of bone marrow
relapse and GVHD | 3-month
  The rate of relapse and GVHD
Event free survival | 1-year
  The rate of event free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, Principal Investigator — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alchalby H, Yunus DR, Zabelina T, Ayuk F, Kroger N. Incidence and risk factors of poor graft function after allogeneic stem cell transplantation for myelofibrosis. Bone Marrow Transplant. 2016 Sep;51(9):1223-7. doi: 10.1038/bmt.2016.98. Epub 2016 Apr 18. PMID 27088376
- [Result] Larocca A, Piaggio G, Podesta M, Pitto A, Bruno B, Di Grazia C, Gualandi F, Occhini D, Raiola AM, Dominietto A, Bregante S, Lamparelli T, Tedone E, Oneto R, Frassoni F, Van Lint MT, Pogliani E, Bacigalupo A. Boost of CD34+-selected peripheral blood cells without further conditioning in patients with poor graft function following allogeneic stem cell transplantation. Haematologica. 2006 Jul;91(7):935-40. PMID 16818281
- [Result] Prabahran A, Koldej R, Chee L, Ritchie D. Clinical features, pathophysiology, and therapy of poor graft function post-allogeneic stem cell transplantation. Blood Adv. 2022 Mar 22;6(6):1947-1959. doi: 10.1182/bloodadvances.2021004537. PMID 34492685
- [Result] Tang Y, Chen J, Liu Q, Chu T, Pan T, Liang J, He XF, Chen F, Yang T, Ma X, Wu X, Hu S, Cao X, Hu X, Hu J, Liu Y, Qi J, Shen Y, Ruan C, Han Y, Wu D. Low-dose decitabine for refractory prolonged isolated thrombocytopenia after HCT: a randomized multicenter trial. Blood Adv. 2021 Mar 9;5(5):1250-1258. doi: 10.1182/bloodadvances.2020002790. PMID 33646303
- [Result] Han Y, Tang Y, Chen J, Liang J, Ye C, Ruan C, Wu D. Low-Dose Decitabine for Patients With Thrombocytopenia Following Allogeneic Hematopoietic Stem Cell Transplantation: A Pilot Therapeutic Study. JAMA Oncol. 2015 May;1(2):249-51. doi: 10.1001/jamaoncol.2014.316. No abstract available. PMID 26181032